CLINICAL TRIAL: NCT01596933
Title: Multi-centric, Placebo-controlled Trial of Omega-3 Fatty Acid Supplementation in Weight Maintenance and Preservation of Lean Body Mass, in (Pre)Cachectic Head and Neck Cancer Patients, Undergoing Curative Radio(Chemo)Therapy
Brief Title: Effect of Omega-3 Supplements on the Prevention of Cachexia in Head and Neck Cancer Treated With Radio(Chemo)Therapy
Acronym: NUTRIOM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: General Hospital Groeninge (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Dr. Philip Debruyne, Consultant Medical Oncologist, General Hospital Groeninge
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NKP_CA_04
Record Dates: First submitted 2012-05-04; First posted 2012-05-11 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Cancer Cachexia; Head and Neck Cancer
Keywords: head and neck cancer; omega-3 fatty acid supplementation; echium oil; weight loss; cancer cachexia; body composition; biomarker; quality of life
MeSH Terms: conditions — Head and Neck Neoplasms; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- omega-3 fatty acid supplementation (Experimental): omega-3 fatty acid supplementation (echium oil)
  Interventions: Dietary Supplement: BioMega SDA®
- standard nutritional support (Placebo Comparator): sunflower oil supplementation
  Interventions: Dietary Supplement: Sunflower oil high oleic

INTERVENTIONS:
Dietary Supplement: BioMega SDA® — Echium oil, 15ml/day, 2 times per oral 7.5ml sachet/day, during 7-week radio(chemo)therapy
  Arms: omega-3 fatty acid supplementation
Dietary Supplement: Sunflower oil high oleic — Sunflower oil high oleic, 15ml/day, 2 times per oral 7.5ml sachet/day, during 7-week radio(chemo)therapy
  Arms: standard nutritional support

SUMMARY:
Cancer cachexia is a complex metabolic process affecting up to 80% of patients suffering from an advanced-stage cancer. Moreover, 20 to 40% of all cancer deaths are caused directly by cachexia. Head and neck (H&N) cancer patients are nutritionally vulnerable since tumour localisation can interfere with food intake, since alcohol and tobacco abuse - two etiological risk factors of H&N cancer - are associated with nutritional deficits, and since the intensive treatment can lead to progressive weight loss. Recently, omega-3 fatty acids have gained interest for their beneficial effects in several diseases. Moreover, nutritional supplementation enriched with omega-3 FA could potentially maintain body weight in cancer patients undergoing intensive treatment.

Aims In this study, the investigators want to evaluate the use of omega-3 FA supplementation as nutritional and the investigators would like to identify potential risk factors, biomarkers and objective measurement tools which can predict therapy-induced cachexia.

DETAILED DESCRIPTION:
Design A prospective, placebo-controlled trial. H&N cancer patients eligible for curative treatment will be randomised to receive standard nutritional support with placebo (15ml/day Sunflower oil, control group) or nutritional support with omega-3 FA supplementation (15ml/day Echium oil, experimental group) during radio(chemo)therapy. All patients will undergo a nutritional screening (Patient-Generated Subjective Global Assessment), a quality of life evaluation (EORTC QLQ C30 & HN35) and will be asked to keep a 3-day food diary at the start of their therapy, and again during the 4th week and the end of therapy. Body composition and grip strength will be measured with bio-electrical impedance (BIA) analysis, Dual X-ray absorptiometry (DXA) and the JAMAR® hydraulic hand dynamometer once at baseline, and again in the 4th week of therapy. Blood samples are collected at baseline, and in the 4th week of therapy to (1) verify compliance rate by measuring fatty acid concentration, (2) verify the presence of potential biomarkers that can predict cachexia and (3) to detect the presence of SNPs associated with severe acute dysphagia. Demographic data, tumour characteristics and therapy-related toxicity will also be collected.

Population Newly diagnosed non-metastatic (stage I-IVB) head and neck cancer patients (≥18 or older) eligible for curative primary or adjuvant radiotherapy with or without systemic therapy

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the head and neck region, generally cancer of the oral cavity, (naso)pharynx and larynx. Cancer of the parotid gland, or nasal cavity and paranasal sinuses are excluded, as well as cT1 N0 M0 tumours of the glottis.
* Primary cancer or relapse, eligible for primary or adjuvant radiotherapy with or without systemic treatment, with curative intent
* TNM stage I to IVB, without distant metastases
* Patients should be older than 18 at the time of enrolment
* Patients should be able to adequately communicate in Dutch or French

Exclusion Criteria:

* Patients younger than 18 years at the time of recruitment
* Pregnant or lactating women
* Patients presenting with another non-cured cancer (PSA or CEA not within normal range as determined by the treating physician)
* Patients that already underwent a radio(chemo)therapy treatment within the last 6 months
* Patients taking oral anticoagulants or LMWH at therapeutic doses
* Patients taking anti-epileptics
* Patients with an indication of heart failure NYHA 3 or 4, or presence of an implantable cardioverter-defibrillator
* Patients with a pacemaker will be excluded from BIA-analysis
* Patients presenting with active intestinal co-morbidity, precluding adequate dietary intake or interfering with the absorption of the nutritional supplements (eg Crohn's disease)
* Patients with a known eating disorder (eg anorexia nervosa, bulimia nervosa)
* Patients with uncontrollable diabetes
* HIV-positive patients
* Patients with (severe) dementia (DSM-IV criteria)
* Patients actively taking fish oil, echium oil or omega-3 FA supplements in the last 4 weeks before enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2012-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
prevention of therapy-related weight loss | 7 weeks
  difference between body weight at baseline and end of therapy

SECONDARY OUTCOMES:
determination of beneficial (and possible side) effects of omega-3 FA supplements in general, and specifically on body weight and body composition | 7 weeks
  measurement of evolution in body composition (baseline - week 4); measurement of evolution in quality of life (baseline - week 4 - end therapy); measurement of adverse events (CTCAE v4.0)in both groups
establish feasibility, variability and distribution of BIA, DXA and JAMAR® as objective measurement tools of body composition | 7 weeks
  evolution percentage fat and lean mass (baseline - week 4) as determined by Bio-Elektrical Impedance (BIA) and Dual Energy X-ray Absorptiometry (DXA); evolution grip strength (kg) (baseline - week 4) as determined by JAMAR® hydraulic hand dynamometer
identification of potential clinical risk factors of cachexia | 7 weeks
  identification of nutritional parameters (obtained from validated nutritional screeners and PG-SGA), demographic, tumour and therapy characteristics, physical, emotional, financial, functional, nutritional and psycho-social characteristics (obtained from EORTC QLQ C30 & HN35), and body composition measurements (% fat, % lean mass, phase angle obtained from BIA, DXA and hand dynamometer)
evaluation of the use and reliability of different validated nutritional screening tools in this population | 7 weeks
  screening with Short Nutritional Assessment Questionnaire (SNAQ), Mini-Nutritional Assessment short-form (MNA-SF), Malnutrition Universal screening tool (MUST), Nutritional risk screening (NRS 2002), Malnutrition screening tool (MST) and the nutrition risk score (NRS); nutritional assessment with Patient Generated - Subjective Global Assessment (PG-SGA) as gold standard
identification and evaluation of potential biomarkers for therapy-induced cachexia | 7 weeks
  identification of serum biomarkers and Single Nucleotide Polymorphisms (SNP)
measurement of difference in quality of life | 7 weeks
  measurement of quality of life (baseline, week 4, end therapy) with EORTC QLQ C30&HN35
dropout and compliance to nutritional supplements | 7 weeks
  number of sachets consumed; omega-3 fatty acid profile as marker for therapy compliance

CONTACTS AND LOCATIONS:
Overall Officials: Philip R Debruyne, MD PhD, Principal Investigator — General Hospital Groeninge; Tom Boterberg, MD PhD, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - Ghent University Hospital, Ghent
  - General Hospital Groeninge, Cancer Center, Kortrijk

REFERENCES:
- [Derived] Pottel L, Lycke M, Boterberg T, Pottel H, Goethals L, Duprez F, Maes A, Goemaere S, Rottey S, Foubert I, Debruyne PR. Echium oil is not protective against weight loss in head and neck cancer patients undergoing curative radio(chemo)therapy: a randomised-controlled trial. BMC Complement Altern Med. 2014 Oct 7;14:382. doi: 10.1186/1472-6882-14-382. PMID 25293388